CLINICAL TRIAL: NCT06142253
Title: Water-based Activity to Enhance Recovery in Long COVID
Brief Title: Water-based Activity to Enhance Recovery in Long COVID-19
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F4647-P
Record Dates: First submitted 2023-11-17; First posted 2023-11-21 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Long COVID
Keywords: Post-Acute COVID-19 Syndrome; Cognitive Training; Exercise; Veterans; Mental Fatigue
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Motor Activity; Mental Fatigue

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomly assigned to one of two groups: 1) Usual Care or 2) WATER+CT
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be blinded to study allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- WATER+CT (Experimental): This is 8-month long two phase intervention consisting of: 1) 6 months of aquatic exercise followed by 2) 2 months of cognitive training.
  Interventions: Behavioral: WATER+CT
- Usual Care (Other): This arm consists of psychoeducation regarding brain health and healthy lifestyles.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: WATER+CT — This is an 8-month long two phase intervention. The first phase consists of 6 months of thrice weekly pool-based exercise occurring at VA Palo Alto. After completion of the 6 month long pool based exercise, participants transition to ten sessions of cognitive training that will occur over 2 months at the VA Palo Alto.
  Arms: WATER+CT
Behavioral: Usual Care — This condition involves receipt of educational materials about brain health and healthy lifestyles as well as regular contact with study staff.
  Arms: Usual Care

SUMMARY:
This two-year study will evaluate the feasibility and safety of an exercise + cognitive training program to improve neurological symptoms of long-COVID. This is a two-phased trial: 1) an exercise phase and 2) a cognitive training phase. The exercise phase will be an aquatic based exercise program. A combination exercise + memory training programs designed for persons with cognitive impairment have significantly improved memory more than other single intervention groups (exercise only, cognitive training only) and given the success of combination training programs with healthy adults, it is important to adapt these programs for persons with neurological symptoms of long-COVID.

DETAILED DESCRIPTION:
The primary research question of the proposed study is this: Is a water-based exercise + cognitive training (WATER+CT) intervention for Veterans with neurological manifestations of long-COVID feasible? The investigators address the need to enhance recovery in this vulnerable population through an innovative multi-component training program that has successfully been used in other cognitively impaired populations. The aims of the proposed research include: 1) demonstrate feasibility as shown by good recruitment and retention rates and stakeholder ratings; 2) evaluate appropriateness of suggested inclusion and exclusion criteria; 3) evaluate acceptability of water-based physical exercise + cognitive training interventions; 4) assess ability of selected outcome measurement techniques to determine the efficacy of water-based physical exercise + cognitive training; and 5) examine outcome "moderator" and "mediator" measurement techniques.

These aims will be tested in a single-blind randomized controlled pilot trial that will establish the feasibility of WATER+CT. This trial will include 50 Veterans, age 18 - 89, experiencing neurological manifestations of long-COVID, with half randomized to WATER+CT and half to usual care. WATER+CT consists of two phases:

1) an exercise training phase and 2) a cognitive training phase. The exercise training (i.e., WATER) consists of a six-month long individualized exercise program of water-based exercises. During this phase, Veterans will come to thrice-weekly group sessions at Aquatic Therapy Center at VA Palo Alto Health Care System (VAPAHCS). After completion of the exercise program, Veterans will begin classroom-based cognitive training at VAPAHCS for up to two months. The CT is based on an efficacious training program that is structured around two components, pre-training, and mnemonic training, both of which have been used successfully in persons with cognitive impairment. Veterans randomized to the UC control condition will receive educational materials about brain health in addition to their usual care, which is the care they would typically receive in the VA. Assessments of adherence will be administered throughout treatment and measures of feasibility will be completed post-treatment.

Participants will complete a variety of neuropsychological measures taping into areas of cognition such as attention, executive functioning, and memory. Participants will also undergo physical fitness assessments including a 6-minute walk test and an exercise treadmill test. To study possible predictors of response to treatment, the investigators will also collect physiological (VO2 max), biological (inflammatory markers and BDNF plasma levels), and genetic data (APOE and BDNF genotypes) from these participants. The investigators hope to provide initial evidence of the feasibility of a water-based exercise training + cognitive training program and provide foundational support for a future program development targeting enhanced recovery in Veterans with neurological manifestations of long-COVID.

ELIGIBILITY:
Inclusion Criteria:

* Veterans, age 18 to 89, of any racial or ethnic group
* Previous COVID-19 infection at least 6 months after diagnosis documented in clinical record
* Persistent neurological symptoms (e.g., "brain fog", cognitive impairment) occurring within 3 months of onset of COVID-19 infection and lasting at least 8 weeks in duration
* Visual and auditory acuity to allow neuropsychological testing
* Willingness to participate in clinical trial for 8 months
* Approval by Primary Care Provider to participate in water-based physical exercise

Exclusion Criteria:

Psychiatric Exclusions

* Current, uncontrolled severe psychotic disorder determined by the Mini International Neuropsychiatric Interview (MINI) Medical Exclusions
* History of neurological (e.g., multiple sclerosis, seizure disorder, stroke,) neurodegenerative (e.g., Parkinson's disease, Alzheimer's disease) or system illness affecting CNS function (e.g., liver failure, kidney failure, congestive heart failure, systemic cancer) occurring before COVID-19 diagnosis
* Current severe cardiac disease (e.g., uncontrolled atrial fibrillation, defined as mean 24 hour heart rate >85 beats/min, or 24 hour maximal ventricular rate >150 beats/min; uncontrolled ventricular arrhythmias, defined as recurrent ventricular tachycardia >3 beats in succession, or 24 hour PVC count >20%; active pericarditis or myocarditis; Class III/IV heart failure and / or ejection fraction < 20%; thrombophlebitis; pulmonary disease with a drop in O2 Sat with exercise to 90% without oxygen; embolism within past 6 months)
* Inability to participate in an exercise stress test
* Inability to read, verbalize understanding and voluntarily sign the Informed Consent

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure | At the end of study completion, an average of 8 months
  The FIM is a brief measure of the feasibility of an intervention.

SECONDARY OUTCOMES:
Acceptability of Intervention Measure | At the end of study completion, an average of 8 months
  The AIM is a brief measure that assesses the acceptability of an intervention.
Change in Fatigue Severity Scale | Through study completion, an average of 8 months
  The Fatigue Severity Scale (FSS) is a method of evaluating the impact of fatigue on a person. The FSS is a short questionnaire that requires a person to rate his/her level of fatigue using a scale of 1 (completely disagree) to 7 (completely agree). Scores range from 9 to 63 with higher scores indicating greater fatigue severity.
Change in Mental Fatigue Scale | Through study completion, an average of 8 months
  The Mental Fatigue Scale (MFS) is self-report scale that includes 15 questions which assess mental fatigue. Items are rated on a scale that ranges from 0 (normal function) to 3 (serious problems). Higher scores indicate greater symptom severity.
Change in Digit Span | Through study completion, an average of 8 months
  The Digit Span subt-test of the WAIS-IV assesses attention and working memory.
Change in Digit Symbol Substitution Test | Through study completion, an average of 8 months
  The Digit Symbol Substitution Test from the WAIS-III assesses attention, processing speed and executive function.
Change in Stroop Color Word Test | Through study completion, an average of 8 months
  The Stroop Color Word test assesses selection attention, cognitive inhibition, and processing speed.
Change in Rey Auditory Verbal Learning Test | Through study completion, an average of 8 months
  The Rey Auditory Verbal Learning Test; (RAVLT) assesses learning and memory.
Change in NIH Toolbox Cognitive Battery | Through study completion, an average of 8 months
  The NIH Toolbox is a computerized battery of test that assesses neuropsychological function.
Change in Hospital Anxiety and Depression Scale | Through study completion, an average of 8 months
  The Hospital Anxiety and Depression Scale (HADS) is a 14-time self-rating scale to assess psychological distress in non-psychiatric patients. Items are rated on a 4-point Likert scale (range 0-3). The total score ranges from 0 to 42 with higher indicating greater severity.
Change in World Health Organization Disability assessment scale 2.0 | Through study completion, an average of 8 months
  The World Health Organization Disability assessment scale 2.0 (WHODAS 2.0) assesses multiple domains of function including: cognition, mobility, self-care, getting along, life activities (household and work) and participation.
Change in Canadian Occupation Performance Measure | Through study completion, an average of 8 months
  The Canadian Occupation Performance Measure (COPM) assesses an individual's perceived occupational performance in the areas of self-care, productivity, and leisure.
Change in Blood labs | Through study completion, an average of 8 months
  Standard blood labs include C-Reactive Protein, Interleukin-6, metabolic panel, and lipid panels
Genetic Testing | Baseline
  Genetic testing includes assessment of APOE and BDNF genotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Kaci Fairchild, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No